CLINICAL TRIAL: NCT03869359
Title: The Effect of Gluten in Patients With Irritable Bowel Syndrome and Healthy Volunteers: a Randomized, Placebo-controlled Double-blind Cross-over Trial
Brief Title: The Effect of Gluten in Patients With Irritable Bowel Syndrome and Healthy Volunteers
Acronym: PROT-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, MD, PhD, Professor, Senior Consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 627-17
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: gluten-free diet; gluten-containing diet; microbiota; metabolomics; healthy volunteers
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Cross-over Trial
Who Masked: Participant, Investigator
Masking Description: The randomization was done by employees of the hospital that were otherwise not involved in the study by drawing concealed envelops. The interventions were concealed plastic bags marked A or B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Gluten-free diet with placebo powder vs Gluten-free diet with gluten powder
  Interventions: Other: Gluten-free diet with gluten powder; Other: Gluten-free diet with placebo powder
- Group B (Experimental): Gluten-free diet with gluten powder vs Gluten-free diet with placebo powder
  Interventions: Other: Gluten-free diet with gluten powder; Other: Gluten-free diet with placebo powder

INTERVENTIONS:
Other: Gluten-free diet with gluten powder — The subjects will sprinkle gluten powder over their meals, twice a day. (14 g/day vital gluten: Real Foods, Edinburgh, United Kingdom). Plastic sachet marked with B (WePack, Derbyshire, United Kingdom). Free of fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs).
Other: Gluten-free diet with placebo powder — The subjects will sprinkle placebo powder over their meals, twice a day. (14 g/day rice starch: Doves Farm Foods Ltd., Berkshire, United Kingdom) Plastic sachets marked with A (WePack, Derbyshire, United Kingdom). Low in fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs).

SUMMARY:
Patients with Irritable Bowel Syndrome (IBS) often link their symptoms to foods. Interest in dietary management recently increased, including the use of a gluten-free diet.

To investigate relation of gluten-free diet (GFD) and IBS, a randomized, double-blind, placebo-controlled cross-over trial will be carried out in adults (>18) and patients with IBS according to Rome IV criteria. The aim is to assess gluten-free versus gluten-containing diet in IBS patients and Healthy Volunteers.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled, cross-over trial.

The aim is to assess the effects of gluten-free diet (GFD) compared to gluten-containing diet (GCD) in IBS patients and Healthy Volunteers on gastrointestinal symptoms, visceral sensitivity, bacterial fermentation, psychological factors and quality of life. The primary hypothesis is that GFD decreases gastrointestinal symptoms compared to GCD and that this change is accompanied with reduced visceral sensitivity and change in bacterial fermentation. The secondary hypothesis is that GFD positively influences psychological factors and quality of life.

IBS patients (Rome IV) and Healthy Volunteers are challenged with gluten in this randomized, double-blind, placebo-controlled, cross-over study. They start with GFD or GCD and cross over to the other intervention (both for 14 days). In between there is a wash-out period of at least 14 days. The subjects will get gluten-free meals (lunch and dinner) and have to sprinkle powder over the meals, concealed in sachets with either gluten (vital gluten) or placebo (rice starch). The subjects will follow a strict GFD during the GFD and GCD periods. The subjects will eat and drink as before the study during the washout period.

Primary outcomes are change in gastrointestinal symptoms, assessed by questionnaires, including IBS Severity Scoring System (IBS-SSS) and Gastrointestinal Symtom Rating Scale-IBS (GSRS-IBS). A 50-point reduction in IBS-SSS indicates clinical response. Bacterial fermentation (exhaled hydrogen and methane) and visceral sensitivity will be measured using the Lactulose-Nutrient Challenge Test. Secondary outcomes are change in psychological factors and quality of life assessed by questionnaires, including CSI, HADS, HSPS, IBSQOL, PHQ-15 and VSI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with IBS according to Rome IV criteria

Exclusion Criteria:

* allergy or documented intolerance to food,
* severe cardiovascular, hepatic, neurological or psychiatric disease
* serious gastrointestinal disease: including celiac disease and inflammatory bowel diseases (IBD),
* diabetes
* bowel dysfunction related to previous surgery
* pregnant or lactating women
* usage of antibiotics within 4 weeks before inclusion
* strict avoidance of foods

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) | Baseline(day 0), day 14, day 28, day 42
  Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) is a validated questionnaire that incorporates typical IBS symptoms such as abdominal pain, abdominal distension and bowel dysfunction, as well as quality of life. Subjects rated their symptoms on a visual analogue scale. The maximum achievable score is 500 points (sum of the 5 scales). A reduction in the total IBS-SSS score of at least 50 points is considered to indicate a clinically significant improvement in symptoms. The scale can also be used to classify IBS symptoms severity: <75 points (no symptoms), 75-175 points (mild symptoms), 175-300 points (moderate symptoms) and >300 points (severe symptoms). Measured after both dietary periods and at baseline of both periods.
Change in Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome (GSRS-IBS) | Baseline(day 0), day 14, day 28, day 42
  Change in Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome (GSRS-IBS) measures symptom severity and symptom frequency in IBS patients and is a reliable and validated questionnaire. Thirteen questions are evaluated and rated from 1 (no discomfort at all) to 7 (very severe discomfort) on a Likert scale. The total scores can range from 13 to 91 (sum of the domains). The GSRS-IBS evaluates 5 domains: abdominal pain, bloating, constipation, diarrhea and satiety. Measured after both dietary periods and at baseline of both periods.
Change in stool frequency, measured by Bristol Stool Form (BSF) | Day 14, Day 42
  Change in Bristol Stool Form, stool frequency per day after both dietary periods
Change in Visceral Sensitivity and Bacterial Fermentation | Baseline(day 0), day 14, day 28, day 42
  Visceral Sensitivity and Bacterial Fermentation measured by the Lactulose-Nutrient Challenge Test.

SECONDARY OUTCOMES:
Change in Central Sensitization Inventory (CSI) score | Baseline(day 0), day 14, day 28, day 42
  The Central Sensitization Inventory (CSI) measures central sensitization related symptoms with 25 questions with a maximum score of 100. A high score indicates high likelihood of central sensitization. Measured after both dietary periods and at baseline of both periods.
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline(day 0), day 14, day 28, day 42
  The Hospital Anxiety and Depression Scale (HADS) contains 7 items for depression and 7 for anxiety. Each item is scored from 0 to 3, and therefore the total score per subscale can range from 0 to 21. When subjects score >10 on 1 or 2 of the subscales, clinically significant psychological distress (anxiety or depression) is likely present. Measured after both dietary periods and at baseline of both periods.
Change in Highly Sensitive Person Scale (HSPS) | Baseline(day 0), day 14, day 28, day 42
  The Highly Sensitive Person Scale (HSPS) contains 27 items and is a valid and reliable questionnaire that measures sensory-processing sensitivity in individuals. Each item is scored from 1 to 7, and therefore the total score can range from 27 to 189. Higher scores indicate high sensory-processing sensitivity. Measured after both dietary periods and at baseline of both periods.
Change in Irritable Bowel Syndrome Quality of Life Questionnaire (IBSQOL) | Baseline(day 0), day 14, day 28, day 42
  The Irritable Bowel Syndrome Quality of Life Questionnaire (IBSQOL) is a 30-item questionnaire that measures quality of life specific to IBS. The IBSQOL is validated and can be used to assess the impact of IBS and possible treatment interventions on quality of life. The following domains are measured: emotional health, mental health, energy, sleep, food/diet, social role, physical functioning, physical role and sexual relations. Scores range from 0 to 100% per domain. Higher scores indicate that IBS influences quality of life greater. Measured after both dietary periods and at baseline of both periods.
Change in Patient health questionnaire-15 (PHQ-15) | Baseline(day 0), day 14, day 28, day 42
  The (PHQ-15) is a validated questionnaire that evaluates 15 somatic symptoms and can be used as a screening tool for somatization in clinical research. The maximum score for men is 28 and 30 for women due to a question about menstrual problems. Measured after both dietary periods and at baseline of both periods.
Change in Visceral Sensitivity Index (VSI) | Baseline(day 0), day 14, day 28, day 42
  The Visceral Sensitivity Index (VSI) is a validated and reliable psychometric instrument which assesses gastrointestinal symptom-specific anxiety. The VSI contains 15 items that are scored from 0 to 5, therefore the total score can range from 0 to 75. Higher scores indicate more severe gastrointestinal symptom-specific anxiety. Measured after both dietary periods and at baseline of both periods.
Change in immunological profile of frozen serum samples | Baseline(day 0), day 14, day 28, day 42
  Frozen serum samples will be analyzed in the future by immunological testing (e.g. ELISA-kit, assays). The future analyses will include interleukins 6 and 8 (IL-6,8) as well as tumor necrosis factor-alpha (TNF-alpha) and immunological markers such as lipopolysaccharide-binding protein (LBP), sCD14, anti-gliadin antibodies (AGA), fibroblast growth factors, fatty acid-binding protein 2, anti-flagellin immunoglobulin G (IgG) and endotoxin-core antibodies immunoglobulin M (IgM). Analyses will be done on samples from before and after both dietary periods.
Change in metabolic profile of frozen urine samples | Baseline(day 0), day 14, day 28, day 42
  Frozen urine samples will be analyzed in the future by metabolome analysis and urine mass spectrometry. For example the metabolites p-hydroxybenzoic acid, histamine and azelaic acid will be measured. Analyses of samples from before and after both dietary periods. Analyses will be done on samples from before and after both dietary periods.
Change in microbiota content of frozen fecal samples | Baseline(day 0), day 14, day 28, day 42
  Fecal microbiota analysis using 16 S RNA technique and Dysbiosis Test. Analyses will be done on samples from before and after both dietary periods.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, MD, PhD, Study Director — Sahlgrenska University Hospital
Locations (1):
- Magnus Simrén, Gothenburg, Västra Götland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Algera JP, Magnusson MK, Ohman L, Storsrud S, Simren M, Tornblom H. Randomised controlled trial: effects of gluten-free diet on symptoms and the gut microenvironment in irritable bowel syndrome. Aliment Pharmacol Ther. 2022 Nov;56(9):1318-1327. doi: 10.1111/apt.17239. Epub 2022 Sep 29. PMID 36173041